CLINICAL TRIAL: NCT05277974
Title: Comparison of Bupivicain Alone With Bupivicain Plus Dexamethasone in Erector Spinae Plane Block For Post-Operative Analgesia After Thoracotomy
Brief Title: Bupivicain vs Bupivicain Plus Dexamethasone in ESP Block for Post-op Analgesia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheikh Zayed Medical College (Other Government)
Responsible Party: Principal Investigator, Amjad Siddique, Assistant Professor, Sheikh Zayed Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASIDDIQUE SZMC
Record Dates: First submitted 2022-03-03; First posted 2022-03-14 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-03

CONDITIONS: Post Operative Pain
Keywords: Erector Spinae Plane Block, Thoracotomy, Ultrasound
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexamethasone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group B. (Active Comparator): group B will receive Inj Bupivicain only in Erector Spinae Plane Block.
  Interventions: Drug: inj bupivicain
- Group D (Active Comparator): group D will receive Inj Bupivicain plus Dexamethasone in Erector Spinae Plane Block.
  Interventions: Drug: inj bupivicain

INTERVENTIONS:
Drug: inj bupivicain — In goup B 30ml of inj. bupivicaine only will be given in Erector Spinae Plane Block and In Group D inj Bupivicain plus inj dexamethasone will be given
  Other Names: inj bupivicain plus dexamethasone

SUMMARY:
Thoracotomy is a very painful procedure. Different treatment modalities are being utilized for post-thoracotomy analgesia including I/V NSAID, Opoids and Neuropathic medications. Other techniques commonly utilized include Thoracic epidural, Paravertebral block; but both are associated with significant failure rate and other complications. Ultrasound guided Erector Spinae Plane block is a new regional anesthesia technique that provides analgesia at multidermatomal levels acriss the posterior, lateral and anterior thoracic walls. The rational of my study is that it is a novel technique and studies with bupivicain alone are present but no study was found with bupivicain plus dexamethasone.

ELIGIBILITY:
Inclusion Criteria:

* age 18-60years ASA I-III Patients undergoing elective thoracotomies

Exclusion Criteria:

* Refusal of Patient Coagulation disorders Known Allergy to Local Anesthetics Infection at the site of injection Pregnant females Morbid Obesity(BMI>40kg/m2) Psychiatric illness Diabetic Patients.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-06-15 (Estimated); Study Completion 2022-07-10 (Estimated)

PRIMARY OUTCOMES:
postoperative pain scores | 36 hours postoperatively
  Visual Analogue Score is utilized to assess the postoperative pain

CONTACTS AND LOCATIONS:
Overall Officials: amjad siddique, FCPS, Principal Investigator — Assistant Professor
Locations (2):
- Pakistan (2):
  - Sheikh Zayed Medical College/Hospital Rahim Yar Khan, Rahim Yar Khan, Punjab Province
  - Sheikh Zayed Medical College/Hospital, Rahim Yar Khan, Punjab Province

IPD SHARING:
Plan to Share IPD: No